CLINICAL TRIAL: NCT01900470
Title: Community Health Worker Support to Help Patients Control Chronic Disease
Brief Title: Effectiveness of Patient-centered Community Health Worker Support to Help Patients Control Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB 817488
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Diabetes; Hypertension; Asthma/COPD With Tobacco Dependence
Keywords: Multiple chronic conditions
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension; Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHW Goal Support (Experimental): IMPaCT CHWs will perform the following functions, depending on the needs of the participants: 1) Deconstructing Distal Goals into Proximal Goals: IMPaCT CHWs will help patients to deconstruct collaborative distal clinical goals into patient driven proximal goals and develop strategies for achieving each proximal goal.2) Creating Roadmaps: Roadmaps are individualized strategies for achieving each proximal goal identified by patients. 3) IMPaCT CHWs conduct weekly follow-up with patients through either telephone or home visit in order to support the achievement of proximal goals. As part of these followup encounters, CHWs ask patients to measure their chronic disease control during their weekly followup calls/visits. 4) Group: CHWs and their Project Manager run a group session for patients in the IMPaCT arm. This group meets weekly and is a forum for patients to discuss common issues around chronic disease management and form a social support network.
  Interventions: Behavioral: CHW Goal Support
- Usual Primary Care (No Intervention): Patients will be encouraged to make follow-up appointments as needed with their primary care clinic for support towards their health goals. During these appointments, clinicians will help patients determine progress made on existing proximal goals, adjust goals based on self-efficacy, and help patients to create new proximal goals as needed. They will also work with PCPs to adjust medications when appropriate, provide health behavior education and make referrals to community-based services based on patient need.

INTERVENTIONS:
Behavioral: CHW Goal Support — IMPaCT CHWs will perform the following functions, depending on the needs of the participants: 1) Deconstructing Distal Goals into Proximal Goals: IMPaCT CHWs will help patients to deconstruct collaborative distal clinical goals into patient driven proximal goals and develop strategies for achieving each proximal goal.2) Creating Roadmaps: Roadmaps are individualized strategies for achieving each proximal goal identified by patients. 3) IMPaCT Partners conduct weekly follow-up with patients through either telephone or home visit in order to support the achievement of proximal goals. As part of these followup encounters, CHWs ask patients to measure their chronic disease control during their weekly followup calls/visits. 4) Group: CHWs and their Project Manager run a group session for patients in the IMPaCT arm. This group meets weekly and is a forum for patients to discuss common issues around chronic disease management and form a social support network.
  Other Names: IMPaCT
  Arms: CHW Goal Support

SUMMARY:
The purpose of this proposal is to compare the effectiveness of community health worker (CHW) support vs. usual primary care for helping chronically-ill, low-SES patients to improve control of chronic conditions. Upon enrollment each patient will select one of their multiple chronic conditions as a focus for the trial and work with his/her PCP to set a chronic disease management goal. Patients are then randomized to receive usual primary care vs. CHW support for moving towards that goal.

ELIGIBILITY:
Inclusion Criteria:

* Patient of target practices for at least 1 yr defined as having one office visit within preceding 12 month
* Home ZIP code including ANY of the following: 1. 19104 2. 19131 3. 19139 4. 19143 5. 19146
* 2 or more of the following conditions: 1. Obesity (BMI greater than 30), 2. HTN (ICD9 relating to HTN in EMR), 3. DM (ICD9 relating to DM in EMR), 4. Asthma/COPD and tobacco dependence (ICD9 for asthma or COPD in EMR AND documentation of tobacco use)
* Uninsured, insured by Medicaid or dually eligible for Medicaid/Managed Medicare
* Patients who have scheduled appointments in the future.

Exclusion Criteria:

* Will not provide informed consent for this study.
* Does not have the capacity to provide informed consent for this study.
* Previously enrolled in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in standardized score | Six months after enrollment
  Six months after enrollment, the IMPaCT arm will have a higher (more negative) mean change in standardized score for chronic disease outcome of interest compared with usual care

SECONDARY OUTCOMES:
Goal achievement | Six months after enrollment
  Six months after enrollment, patients in the IMPaCT group will have higher proportion of patients who achieve their individualized chronic disease management goal compared with usual care
SF-12 | Six months after enrollment,
  Six months after enrollment, patients in the IMPaCT group will greater improvements in their self-rated health (as measured by mean change in MCS and PCS of the SF-12) than patients receiving usual care.
CAHPS PCMH (Communication, Self-Management Support, Comprehensiveness of Care) | Six months after enrollment
  Six months after enrollment, the IMPaCT arm will have higher perceived quality of patient-centered medical care (as measured by the Consumer Assessment of Healthcare Providers and Systems Patient-Centered Medical Home (CAHPS PCMH) survey) than the usual care arm. Specifically, we will measure the CAHPS PCMH domains pertaining to Self-Management Support and Comprehensiveness of Care.
Hospitalization | 6 months after enrollment
  Patients in the IMpaCT arm with have a lower rate of hospitalizations than the usual care arm at 6 months after enrollment.
Patient Activation | Six months after enrollment
  Six months after enrollment, patients in the IMPaCT arm will have greater improvements in their activation (as measured by mean change in PAM score) compared with patients in the usual care arm.

OTHER OUTCOMES:
Hospitalizations at 12 months | 12 months after enrollment
  Patients in the IMpaCT arm with have a lower rate of hospitalizations than the usual care arm at 12 months after enrollment.
Medical Adherence | Six months after enrollment
  Six months after enrollment, patients in the IMPaCT arm will have higher levels of adherence to medical recommendations than the usual care arm, as measured by the Medical Outcomes Study (MOS) Measures of Patient Adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Shreya Kangovi, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kangovi S, Mitra N, Grande D, Huo H, Smith RA, Long JA. Community Health Worker Support for Disadvantaged Patients With Multiple Chronic Diseases: A Randomized Clinical Trial. Am J Public Health. 2017 Oct;107(10):1660-1667. doi: 10.2105/AJPH.2017.303985. Epub 2017 Aug 17. PMID 28817334
- [Derived] Kangovi S, Mitra N, Turr L, Huo H, Grande D, Long JA. A randomized controlled trial of a community health worker intervention in a population of patients with multiple chronic diseases: Study design and protocol. Contemp Clin Trials. 2017 Feb;53:115-121. doi: 10.1016/j.cct.2016.12.009. Epub 2016 Dec 10. PMID 27965180
- [Derived] Kangovi S, Mitra N, Smith RA, Kulkarni R, Turr L, Huo H, Glanz K, Grande D, Long JA. Decision-making and goal-setting in chronic disease management: Baseline findings of a randomized controlled trial. Patient Educ Couns. 2017 Mar;100(3):449-455. doi: 10.1016/j.pec.2016.09.019. Epub 2016 Sep 25. PMID 27717532